CLINICAL TRIAL: NCT02308124
Title: Treatment and Prognosis of Neurogenic Orthostatic Hypotension : A Prospective Randomized Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kon Chu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1409066609
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Orthostatic; Hypotension, Neurogenic
MeSH Terms: conditions — Hypotension | interventions — Midodrine; Pyridostigmine Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Midodrine (Experimental): Start midodrine 2.5mg bid, and then dose up to 5mg bid after one month if necessary.
  Interventions: Drug: Midodrine
- Pyridostigmine (Experimental): Start Pyridostigmine 30mg bid, and then dose up to 60mg bid after one month if necessary.
  Interventions: Drug: Pyridostigmine Bromide
- Midodrine + Pyridostigmine (Experimental): Start midodrine 2.5mg bid+ Pyridostigmine 30mg bid, and then dose up to midodrine 5mg bid+ Pyridostigmine 60mg bid after one month if necessary.
  Interventions: Drug: Midodrine + pyridostigmine

INTERVENTIONS:
Drug: Midodrine
  Other Names: Midodrine only
  Arms: Midodrine
Drug: Pyridostigmine Bromide
  Other Names: Pyridostigmine only
  Arms: Pyridostigmine
Drug: Midodrine + pyridostigmine
  Other Names: Combination
  Arms: Midodrine + Pyridostigmine

SUMMARY:
Compare the effect of treatment of midodrine and pyridostigmine in neurogenic orthostatic hypotension and investigate the quality of life of treatment of neurogenic orthostatic hypotension.

DETAILED DESCRIPTION:
In patients with neurogenic orthostatic hypotension, the appropriate treatment was identified by comparing the treatment effects and side effects for each treatment drug. In addition, by confirming the effect of orthostatic hypotension on lowering the quality of life, it is expected that the improvement of the quality of life will help.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 patients who complained of dizziness
* Orthostatic hypotension after 3-minute standing (systolic blood pressure drop >=20 or diastolic blood pressure drop >=10

Exclusion Criteria:

* Drug-induced hypotension, if necessary, evaluate patient after discontinuing the causative drug for one month
* Heart failure or Chronic renal failure
* Patients who cannot or do not want to write questionaires.
* Poor drug compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kon Chu, Principal Investigator — Seoul National University Hospital, Seoul, South Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Arbique D, Cheek D, Welliver M, Vongpatanasin W. Management of neurogenic orthostatic hypotension. J Am Med Dir Assoc. 2014 Apr;15(4):234-9. doi: 10.1016/j.jamda.2013.10.014. Epub 2014 Jan 2. PMID 24388946
- [Background] Smith ND. Orthostatic Hypotension in the Patient with Diabetes: A Broad Review of Pharmacologic Treatment Options. Journal of Pharmacy Technology. 2013 January 1, 2013;29(1):23-34.
- [Background] Low PA, Singer W. Management of neurogenic orthostatic hypotension: an update. Lancet Neurol. 2008 May;7(5):451-8. doi: 10.1016/S1474-4422(08)70088-7. PMID 18420158
- [Background] Shibao C, Grijalva CG, Raj SR, Biaggioni I, Griffin MR. Orthostatic hypotension-related hospitalizations in the United States. Am J Med. 2007 Nov;120(11):975-80. doi: 10.1016/j.amjmed.2007.05.009. PMID 17976425
- [Background] Goldstein DS, Sharabi Y. Neurogenic orthostatic hypotension: a pathophysiological approach. Circulation. 2009 Jan 6;119(1):139-46. doi: 10.1161/CIRCULATIONAHA.108.805887. No abstract available. PMID 19124673
- [Background] Lahrmann H, Cortelli P, Hilz M, Mathias CJ, Struhal W, Tassinari M. EFNS guidelines on the diagnosis and management of orthostatic hypotension. Eur J Neurol. 2006 Sep;13(9):930-6. doi: 10.1111/j.1468-1331.2006.01512.x. PMID 16930356
- [Background] Parsaik AK, Singh B, Altayar O, Mascarenhas SS, Singh SK, Erwin PJ, Murad MH. Midodrine for orthostatic hypotension: a systematic review and meta-analysis of clinical trials. J Gen Intern Med. 2013 Nov;28(11):1496-503. doi: 10.1007/s11606-013-2520-3. Epub 2013 Jun 18. PMID 23775146
- [Background] Wright RA, Kaufmann HC, Perera R, Opfer-Gehrking TL, McElligott MA, Sheng KN, Low PA. A double-blind, dose-response study of midodrine in neurogenic orthostatic hypotension. Neurology. 1998 Jul;51(1):120-4. doi: 10.1212/wnl.51.1.120. PMID 9674789
- [Background] Kaufmann H, Malamut R, Norcliffe-Kaufmann L, Rosa K, Freeman R. The Orthostatic Hypotension Questionnaire (OHQ): validation of a novel symptom assessment scale. Clin Auton Res. 2012 Apr;22(2):79-90. doi: 10.1007/s10286-011-0146-2. Epub 2011 Nov 2. PMID 22045363
- [Background] Jankovic J, Gilden JL, Hiner BC, Kaufmann H, Brown DC, Coghlan CH, Rubin M, Fouad-Tarazi FM. Neurogenic orthostatic hypotension: a double-blind, placebo-controlled study with midodrine. Am J Med. 1993 Jul;95(1):38-48. doi: 10.1016/0002-9343(93)90230-m. PMID 7687093
- [Background] Low PA, Gilden JL, Freeman R, Sheng KN, McElligott MA. Efficacy of midodrine vs placebo in neurogenic orthostatic hypotension. A randomized, double-blind multicenter study. Midodrine Study Group. JAMA. 1997 Apr 2;277(13):1046-51. PMID 9091692
- [Background] Singer W, Opfer-Gehrking TL, McPhee BR, Hilz MJ, Bharucha AE, Low PA. Acetylcholinesterase inhibition: a novel approach in the treatment of neurogenic orthostatic hypotension. J Neurol Neurosurg Psychiatry. 2003 Sep;74(9):1294-8. doi: 10.1136/jnnp.74.9.1294. PMID 12933939
- [Background] Singer W, Sandroni P, Opfer-Gehrking TL, Suarez GA, Klein CM, Hines S, O'Brien PC, Slezak J, Low PA. Pyridostigmine treatment trial in neurogenic orthostatic hypotension. Arch Neurol. 2006 Apr;63(4):513-8. doi: 10.1001/archneur.63.4.noc50340. Epub 2006 Feb 13. PMID 16476804
- [Derived] Byun JI, Moon J, Kim DY, Shin H, Sunwoo JS, Lim JA, Kim TJ, Lee WJ, Lee HS, Jun JS, Park KI, Lee ST, Jung KH, Jung KY, Lee SK, Chu K. Efficacy of single or combined midodrine and pyridostigmine in orthostatic hypotension. Neurology. 2017 Sep 5;89(10):1078-1086. doi: 10.1212/WNL.0000000000004340. Epub 2017 Aug 9. PMID 28794253

RESULTS

PARTICIPANT FLOW:
Groups:
- Midodrine Only: Start midodrine 2.5mg bid, and then dose up to 5mg bid after one month if necessary.
- Pyridostigmine Only: Start Pyridostigmine 30mg bid, and then dose up to 60mg bid after one month if necessary.
Period: Overall Study
Arm/Group | Midodrine Only | Pyridostigmine Only | Midodrine + Pyridostigmine
Started | 29 | 29 | 29
Completed | 23 | 21 | 21
Not Completed | 6 | 8 | 8
Not completed — Lost to Follow-up | 6 | 6 | 6
Not completed — Adverse Event | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midodrine Only | Pyridostigmine Only | Midodrine + Pyridostigmine | Total
Number analyzed (Participants) | 29 | 29 | 29 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (17.7) | 59.7 (13.4) | 52.7 (16.2) | 57.2 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 15 | 46
  Male | 15 | 12 | 14 | 41
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 29 | 29 | 29 | 87
Supine systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 137.3 (20.9) | 124.5 (18.5) | 122.0 (15.6) | 127.9 (19.4)
Supine diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 83.2 (12.8) | 76.5 (9.8) | 76.9 (10.4) | 78.9 (11.4)
Supine heart rate [Mean (Standard Deviation); unit: Beats per Minute] | 68.0 (11.3) | 66.7 (13.5) | 67.0 (10.7) | 67.2 (11.8)
Orthostatic systolic blood pressure change [Mean (Standard Deviation); unit: mmHg] — Maximum decrements in SBP within 3 minutes of standing were recorded.
  mmHg | -24.7 (9.9) | -23.3 (12.5) | -22.5 (10.1) | -23.5 (10.8)
Orthostatic diastolic blood pressure change [Mean (Standard Deviation); unit: mmHg] — Maximum decrements in DBP within 3 minutes of standing were recorded.
  mmHg | -13.4 (9.0) | -15.5 (9.9) | -13.4 (8.2) | -14.1 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Orthostatic BP Drop
Description: Change of orthostatic SBP and DBP drop after 3-month medical treatment compared to initial results.
Time Frame: after 3-month medical treatment
Population: At 3 months after treatment, 65 patients were evaluated (Midodrine only; 23, Pyridostigmine only; 21, Midodrine + Pyridostigmine; 21). 22 additional patients missed visit (Midodrine only; 6, Pyridostigmine only; 8, Midodrine + Pyridostigmine; 8)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Midodrine Only | Pyridostigmine Only | Midodrine + Pyridostigmine
Number analyzed (Participants) | 23 | 21 | 21
mmHg
  Changes in SBP drop | 11.1 (16.9) | 13.6 (20.1) | 8.9 (9.9)
  Changes in DBP drop | 7.5 (15.3) | 11.1 (17.7) | 7.4 (14.2)

2. Secondary Outcome: Change of the Orthostatic Hypotension Associated Symptom Questionnaire (OH Questionnaire (OHQ)).
Description: Change of the OH associated symptom survey result after 3-month medical treatment compared to initial results.
  OHQ questionnaire has two components: the OH daily activity scale (OHDAS), which contains 4 items measuring the impact of OH on daily activities, and the OH symptom assessment (OHSA), which contains 6 items measuring the symptoms of OH (dizziness/light headedness, vision disturbance, weakness, fatigue, trouble concentrating, and head/neck discomfort).This questionnaire reflects the severity of OH-related symptoms on a 10-point scale, with 0 indicating the absence of a symptom and 10 indicating maximal severity.
  ** OHQ total score minimal 0 ~ maximal 100
Time Frame: after 3-month medical treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Midodrine Only | Pyridostigmine Only | Midodrine + Pyridostigmine
Number analyzed (Participants) | 23 | 21 | 21
points | -16.2 (15.5) | -17.2 (20.3) | -12.6 (14.8)

3. Secondary Outcome: Change of the Depression Score (Beck Depression Inventory-II )
Description: Change of the depression score after 3-month medical treatment compared to initial results.
  21 multiple-choice questions, each of which can be scored from 0 to 3. Higher score represent higher degree of depression.
  Score Normal; 0-13, Mild depression; 14-19, Moderate depression; 20-28, Severe depression; 29-63
Time Frame: after 3-month medical treatment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Midodrine Only | Pyridostigmine Only | Midodrine + Pyridostigmine
Number analyzed (Participants) | 23 | 21 | 21
points | -6.8 (5.6) | -7.8 (6.5) | -3.5 (8.0)

4. Secondary Outcome: Short-form 36 Version 2
Description: changes in Short Form (36) Health Survey version 2 (SF-36v2) physical component summary scale (PCS) compared to the baseline
  SF-36v2 measures eight HRQOL domains (physical functioning, role limitation caused by physical problems, bodily pain, general health, vitality, social functioning, role limitation caused by emotional problems, and mental health) summarized into two summary scales that are normalized to the population (mean=50, standard deviation=10): the physical component summary scale (PCS) and the mental component summary scale (MCS).20 Better HRQOL is reflected by higher SF-36v2 scores.
Time Frame: changes at 3 months after treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Midodrine Only | Pyridostigmine Only | Midodrine + Pyridostigmine
Number analyzed (Participants) | 23 | 21 | 21
points | 5.6 (6.8) | 4.2 (9.1) | 2.7 (7.0)

5. Secondary Outcome: Changes in Health-related Quality of Life
Description: changes in Short Form (36) Health Survey version 2 (SF-36v2) mental component summary scale (MCS)
  SF-36v2 measures eight HRQOL domains (physical functioning, role limitation caused by physical problems, bodily pain, general health, vitality, social functioning, role limitation caused by emotional problems, and mental health) summarized into two summary scales that are normalized to the population (mean=50, standard deviation=10): the physical component summary scale (PCS) and the mental component summary scale (MCS).20 Better HRQOL is reflected by higher SF-36v2 scores.
Time Frame: changes at 3 months after treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Midodrine Only | Pyridostigmine Only | Midodrine + Pyridostigmine
Number analyzed (Participants) | 23 | 21 | 21
points | 5.0 (8.6) | 6.7 (8.9) | 0.4 (11.2)

ADVERSE EVENTS:
Time Frame: Possible side effects were checked by direct questioning at each visit at 1 and 3 months after treatment. Expected adverse reactions were listed in the protocol.
Arm/Group | Midodrine Only | Pyridostigmine Only | Midodrine + Pyridostigmine
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 1/29 | 6/29 | 3/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midodrine Only (N=29) | Pyridostigmine Only (N=29) | Midodrine + Pyridostigmine (N=29)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study lacked a placebo group and a blinding process Compared with previous studies, which focused on primary autonomic degenerative disorders, our study included more patients with peripheral autonomic neuropathy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No